CLINICAL TRIAL: NCT01400880
Title: Electrode-based Sensor for Non-invasive Fetal Heart Rate and EMG Monitoring With Improved Reliability
Status: Completed | Type: Observational
Sponsor: Convergent Engineering, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: Conveng-001
Record Dates: First submitted 2011-07-21; First posted 2011-07-22 (Estimated); Results first posted 2015-02-12 (Estimated); Last update posted 2015-02-12 (Estimated); Status verified 2015-02

CONDITIONS: Pregnancy
Keywords: Maternal Fetal Monitoring

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pregnant: In Labor

SUMMARY:
The specific goal of the proposed research is to develop a reliable, non-invasive fetal and maternal heart rate and contraction monitor that is unaffected by obesity and requires less nursing intervention than the tocodynamometer and Doppler ultrasound.

DETAILED DESCRIPTION:
The majority of obstetric deliveries in the US undergo electronic monitoring and continuous uterine activity and fetal heart rate (FHR) monitoring is the standard of care. Typically, external transducers are employed, the reliability of which depends on their proper positioning, which may be disturbed by patient or fetal movement. The tocodynamometer (strain gauge, toco for short) provides frequency and timing of contractions, but requires transmission of tension from the uterus to the sensor. Fetal heart rate is acquired with an external Doppler ultrasound transducer. The reliability of this monitor depends on the ability to obtain a window to the fetal heart.

In some patients, particularly the obese, the toco and ultrasound may fail to monitor consistently. In others both transducers require frequent repositioning by the nursing staff, and the Doppler may erroneously report maternal heart rate instead of fetal.

The alternative uterine activity monitor is an intrauterine pressure catheter (IUPC), which is placed through the cervical os in the adequately dilated patient with ruptured membranes. While this monitor usually provides a more reliable signal than the toco, as well as quantitative information regarding intrauterine pressure, it is invasive and there is an increased risk of infection. The alternative FHR monitor is via fetal scalp electrode (FSE), which is applied transvaginally to the fetal presenting part, also requiring adequate cervical dilation and ruptured membranes. While the FSE usually provides a more reliable signal, it is similarly invasive and increases risk of infection.

ELIGIBILITY:
Inclusion Criteria:

* Women between the ages of 18 and 50 years old
* >/= 34 weeks gestation
* Single viable fetus in cephalic presentation

Exclusion Criteria:

* Bleeding or uterine scarring

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Laboring women in Labor and Delivery ward
Sampling Method: Non-Probability Sample
Enrollment: 103 (Actual)
Dates: Start 2011-07; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Gregg, PhD, Principal Investigator — University of Florida
Locations (1):
- University of Florida College of Medicine, Gainesville, Florida, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Electrode Sensor, TOCO and IUPC: Pregnant women between the ages of 18-50 with a single viable fetus in cephalic presentation monitored with Electrode Sensor, TOCO and IUPC
Period: Overall Study
Arm/Group | Electrode Sensor, TOCO and IUPC
Started | 103 (patients were added throughout the study. There was not a set number of patients that we began with)
Completed | 101 (patients were added throughout the study. There was not a set number of patients that we began with)
Not Completed | 2

BASELINE CHARACTERISTICS:
Population: The number of participants was determined by the time allowable by the IRB approval for the site study.
Groups:
- Primary: Pregnant women between the ages of 18-50 with a single viable fetus in cephalic presentation
Arm/Group | Primary
Number analyzed (Participants) | 101
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 101
  >=65 years | 0
Sex/Gender, Customized [Number; unit: participants]
  Pregnant Women | 101

OUTCOME MEASURES:

1. Primary Outcome: Comparison of Electrode Sensor and TOCO Detection of Contraction Events, as Compared to IUPC
Description: Contraction timing as measured by the electrode sensor and contraction timing as measure by the TOCO, both compared to the contraction timing as measured by the IUPC gold standard. The contraction timing values of the electrode sensor and TOCO were then compared.
Time Frame: Stage I and II Labor
Population: Pregnant women between the ages of 18-50 with a single viable fetus in stages I and/or II of labor
Measure: Mean (Standard Deviation); unit: seconds
Groups:
- Electrode Sensor, TOCO and IUPC: Pregnant women between the ages of 18-50 with a single viable fetus in cephalic presentation studied with electrode sensor, Tocodynamometer and IUPC
Arm/Group | Electrode Sensor, TOCO and IUPC
Number analyzed (Participants) | 101
seconds
  TOCO patient group | 2.98 (3.28)
  Electrode Sensor patient group | 3.95 (2.65)
Statistical Analysis 1: Comparison: Electrode Sensor, TOCO and IUPC; All subjects were monitored with the electrode sensor, TOCO and IUPC. Measurements were taken with the electrode sensor vs. IUPC and were also taken with TOCO vs. IUPC and those measurements were compared to each other. These results are for TOCO and IUPC. Agreement between TOCO and IUPC. Null hypothesis: the mean peak difference between TOCO and IUPC is equal to 0. Alternative hypothesis: the mean peak difference is not equal to 0; Test type: Superiority or Other; Mean Difference (Final Values) = 2.98, 95% CI 2-sided [1.70 to 4.27], Standard Deviation 3.28
Statistical Analysis 2: Comparison: Electrode Sensor, TOCO and IUPC; All subjects were monitored with the electrode sensor, TOCO and IUPC. Measurements were taken with the electrode sensor vs. IUPC and were also taken with TOCO vs. IUPC and those measurements were compared to each other. These results are for the electrode sensor and IUPC. Agreement between electrode sensor and IUPC. Null hypothesis: the mean peak difference between TOCO and IUPC is equal to 0. Alternative hypothesis: the mean peak difference is not equal to 0; Test type: Superiority or Other; Mean Difference (Final Values) = 3.95, 95% CI 2-sided [2.98 to 4.92], Standard Deviation 2.65

ADVERSE EVENTS:
Time Frame: Adverse events occurred throughout the study dates starting 8/1/11 and ending 4/25/13. 1 year 9 months.
Description: All adverse events were recorded, even if the event was not directly related to the study. Some patients developed infection directly after data collection started and thus were already infected, not being caused by the study. Also, C-sections were reported as it disrupted the data collection and was not a foreseeable event.
Arm/Group | Primary
Serious Adverse Events (participants affected / at risk) | 0/103
Other Adverse Events (participants affected / at risk) | 15/103
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Primary (N=103)
Chorioamnionitis (Infections and infestations) | 13 (13) — Patient developed Chorioamnionitis after IUPC, electrodes and toco were placed either for OB monitoring or study reasons. All patients were treated and infection resolved. Infection unlikely a result of study, but cannot be ruled out.
c-section (Surgical and medical procedures) | 2 (2) — Patients were prepped for C-section deliveries and thus data collection was discontinued. These were not related to the study data collection. Doctor felt fetus needed to be delivered.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No